CLINICAL TRIAL: NCT05845567
Title: An Open-label, Single-center, Study in Healthy Subjects to Investigate the Effect of Oral Clarithromycin on the Pharmacokinetics of Givinostat (PART 2)
Brief Title: The Potential of Givinostat as DDI Victim in Co-administration P-gp Inhibitor (Part 2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITF/2357/55 - PART 2; 2021-005756-11 (EudraCT Number)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-07

CONDITIONS: Drug Drug Interaction
Keywords: PK; Pharmacokinetics; Givinostat; Clarythromycin
MeSH Terms: interventions — givinostat; givinostat hydrochloride; Clarithromycin

STUDY DESIGN:
Masking Description: The study was conducted as open label. Blinding procedures were not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Givinostat + Clarithromycin (Experimental): Givinostat and Clarithromycin Days 1 and 8, Givinostat 50 mg as oral suspension was administered as a single dose, 1 hour after Clarithromycin administration. From Day 4 to Day 10, Clarithromycin 500 mg film-coated tablet was administered twice a day.
  Interventions: Drug: Givinostat; Drug: Clarithromycin

INTERVENTIONS:
Drug: Givinostat — ITF2357 Givinostat 10mg/mL. Dose: 10 mg/mL; Dosage form: oral suspension.
  Other Names: ITF2357
Drug: Clarithromycin — Clarithromycin 500 mg immediate-release oral film-coated tablet (Klacid®) was administered twice a day, in the morning and in the evening.
  Other Names: Klacid®

SUMMARY:
Primary objective:

To assess the potential effect of oral Clarithromycin on the single-dose pharmacokinetics of Givinostat.

Secondary objective:

To assess the safety and tolerability of concomitant administration of Givinostat plus Clarithromycin.

DETAILED DESCRIPTION:
This study was planned as a phase I, open-label, 3-part, fixed-sequence, non-randomized study in healthy male and female subjects. The study (Part 2) aimed at assessing the potential effect of Clarythromycin on the single dose pharmacokynetics of Givinostat.

The total duration of Part 2 was divided as follows:

* Screening: up to 21 days.
* Treatment Period: Days 1 to 11.
* Safety follow-up visit: 12±2 days.

Subjects were confined at site from Day -1 to Day 11. On Days 1 and 8, a single dose of 50 mg Givinostat, as oral suspension, was administered 1 hour after the planned morning time of Clarithromycin administration.

From Day 4 to Day 10, clarithromycin 500 mg film-coated tablets were administered twice a day, in the morning and in the evening.

The following assessments were performed:

* Blood collection for pharmacokinetic analysis on Days 1 to 4 and 8 to 11.
* Vital signs measurements on Days 1 and 4 to 10.
* 12-lead ECG on Days 1, 3, 7 and 8.
* Blood collection for laboratory tests (hematology and biochemistry) on Day 3.

Subjects were discharged in the morning of Day 11 after completing end of study procedures.

ELIGIBILITY:
Inclusion Criteria:

* A subject was considered eligible for the study if he/she fulfilled all the inclusion criteria:

  1. Subject's written informed consent obtained prior to any study-related procedure.
  2. Male or female subject, ≥18 and ≤55 years of age, at the time of signing the informed consent.
  3. Body mass index (BMI) of 18.5 to 32.0 kg/m2 inclusive, and body weight ≥55 kg and ≤100 kg for females and body weight ≥60 kg and ≤110 kg for males.
  4. Non-smoker or ex-smoker (i.e. someone who abstained from using tobacco or nicotine-containing products for at least 3 months prior to Screening).
  5. No clinically relevant diseases.
  6. No major surgery within 4 weeks prior to dosing.
  7. No clinically relevant abnormalities on physical examination.
  8. No clinically relevant abnormalities on 12-lead ECG.
  9. No clinically relevant abnormalities on clinical laboratory tests.
  10. Negative test results for anti-Human Immunodeficiency virus 1 and 2 antibodies (anti-HIV-1Ab and anti-HIV-2Ab), Hepatitis B surface antigen (HBsAg) and anti-Hepatitis C virus antibodies (anti-HCVAb).
  11. Female subjects are eligible if they are of non-childbearing potential or agree to use a non-hormonal highly effective contraceptive method from 28 days prior to Screening until at least 90 days after the last study drug administration. Nonchildbearing potential female is defined as:

      1. Menopausal, i.e. no menses for ≥ 12 months without an alternative medical cause other than menopause, and a high FSH level.
      2. Pre-menopausal female with documented hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy.

      A non-hormonal effective contraceptive method is defined as:
      1. Intrauterine device.
      2. Bilateral tubal occlusion.
      3. Total abstinence of heterosexual intercourse, in accordance with the lifestyle of the subject.
      4. Vasectomized partner, who has received medical assessment of the surgical success, or clinically diagnosed infertile partner.
  12. Male subjects who are sexually active with a female partner of childbearing potential (pregnant or non-pregnant) must use contraception (condom) from investigational product administration up to at least 90 days following the last study drug administration.
  13. Male subjects must ensure that his non-pregnant female partner of childbearing potential agrees to consistently and correctly use for the same period a highly effective method of contraception (see Section 8.5.3).
  14. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
  15. Willingness and capability to comply with the requirements of the study and ability to understand the study procedures and the risks involved.

      Exclusion Criteria
* A subject was excluded from the study if he/she fulfilled any of the exclusion criteria:

At Screening

1. Previous use of Givinostat.
2. History of anaphylaxis reaction or clinically significant drug hypersensitivity reaction (e.g., angioedema, Stevens-Johnson syndrome, acute generalized exanthematous pustulosis, drug-induced hypersensitivity syndrome, druginduced neutropenia).
3. Known history of hypersensitivity and/or allergic reactions to Givinostat, histone deacetylases (HDAC) inhibitors or to any excipient in the formulation.
4. History of sorbitol intolerance, sorbitol malabsorption or fructose intolerance.
5. Any medical condition (e.g. gastrointestinal, renal or hepatic, including peptic ulcer, inflammatory bowel disease or pancreatitis) or surgical condition (e.g. cholecystectomy, gastrectomy) that may affect drug pharmacokinetics (absorption, distribution, metabolism or excretion) or subject safety.
6. Systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg, or pulse rate lower than 50 or over 100 bpm.
7. QTcF ˃450 msec.
8. Subjects with history of cardiac arrhythmias (documented), family history of sudden cardiac death or history of additional risk factors for torsades-depointes (e.g. heart failure, hypokalemia, long QT syndrome).
9. Having an estimated glomerular filtration (eGFR) < 90 mL/min, based on creatinine clearance calculation by the Cockcroft-Gault formula and normalized to an average surface area of 1.73 m2.
10. Any of the following abnormal laboratory test values:

    1. Platelet count below the lower limit of the normal range (LLN).
    2. Total white blood cells count below the LLN.
    3. Hemoglobin below the LLN.
    4. Triglycerides above the upper limit of normal range (ULN).
    5. Potassium or magnesium below the LLN.
11. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
12. Positive serum pregnancy test.
13. If woman, she is breast-feeding.
14. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (i.e. more than 14 units of alcohol per week for males or more than 7 units for females).
15. History of drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs [such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives] within 1 year prior to screening.
16. Participation in any clinical trial within the previous 2 months.
17. Participation in more than 2 clinical trials within the previous 12 months.
18. Blood donation or significant blood loss (≥ 450 mL) due to any reason or had plasmapheresis within the previous 2 months.
19. Veins unsuitable for intravenous puncture on either arm.
20. Difficulty in swallowing capsules, tablets or suspensions.
21. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
22. Known history of hypersensitivity and/or allergic reactions to clarithromycin, other macrolides or to any excipient in the formulation.

    At Admission to Treatment Period
23. Any clinically relevant abnormalities on clinical laboratory tests.
24. Positive urine alcohol, drugs-of-abuse or cotinine screen tests.
25. Positive urine pregnancy test.
26. Positive or inconclusive SARS-CoV-2 test prior to admission.
27. Use of prescription or non-prescription medicinal products within the previous 28 days or within 5-half-lives of the medicinal product, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Fonseca, MD, Principal Investigator — Blueclinical, Ltd.
Locations (1):
- Hospital da Prelada, 3rd Floor & East Wing 4th Floor Rua Sarmento de Beires, Porto, Portugal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients were enrolled. One discontinued after first dosing, so while safety and PK analysis populations were composed of 20 subjects, the drug-drug interaction comparable bioavailability is calculated on 19 subjects.
Groups:
- Total Subjects Enrolled: At Day 1 patients received Givinostat 50 mg. At Days 4-7 patients received Clarithromycin 500 mg b.i.d. At Day 8 patients received Givinostat 50 mg + Clarithromycin 500 mg b.i.d At Days 9-10 patients received Clarithromycin 500 mg b.i.d.
  Givinostat: ITF2357 Givinostat 10mg/mL. Dose: 10 mg/mL; Dosage form: oral suspension.
  Clarithromycin: Clarithromycin 500 mg immediate-release oral film-coated tablet (Klacid®) administered twice a day, in the morning and in the evening.
Period: Overall Study
Arm/Group | Total Subjects Enrolled
Started | 20
Safety Analysis Population | 20
PK Analysis Population | 20
Drug-Drug Interaction Comparable Bioavailability | 19
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Twenty (20) subjects received at least one dose of an IMP in the study. They constitute the Safety Analysis Population.
Arm/Group | Total Subjects Enrolled
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Portugal | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Givinostat, Following Single Doses of the Parent Drug
Description: Maximum observed plasma concentration (Cmax) of givinostat.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of Givinostat.
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: Pharmacokinetic Analysis Population: subjects enrolled in the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation.
  Please note that one of the 20 PK subjects early withdrew from the study before taking any study drug. This explains why patients analyzed in the combo arm are n=19 and not n=20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Givinostat Alone (Day 1): Givinostat 10 mg/mL oral suspension was administered as a single dose, alone, on Day 1.
- Givinostat Co-Administered With Clarithromycin (Day 8): Givinostat 10 mg/mL oral suspension was administered as a single dose, in combination with Clarithromycin 500 mg immediate-release film-coated tablets (Klacid®) on Day 8.
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 20 | 19
ng/mL | 53.57 (24.2) | 75.35 (21.9)
Statistical Analysis 1: Comparison: Givinostat Alone (Day 1) vs Givinostat Co-Administered With Clarithromycin (Day 8); Test type: Superiority; ratio of the Geometric LSmeans = 139.43, 90% CI 2-sided [129.73 to 149.86]

2. Primary Outcome: AUC0-t of Givinostat, Following Single Doses of the Parent Drug
Description: AUC0-t = area under the curve from time zero to last sampling time with quantifiable concentrations.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of Givinostat, on Days 1 and 8, for the determination of Givinostat.
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: Pharmacokinetic Analysis Population: subjects enrolled in the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation. Please note that one of the 20 PK subjects early withdrew from the study before taking any study drug. Please note that one of the 20 PK subjects early withdrew from the study before taking any study drug. This explains why patients analyzed in each arm are n=19 and not n=20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 19 | 19
ng.h/mL | 344.67 (20.4) | 406.61 (13.0)
Statistical Analysis 1: Comparison: Givinostat Alone (Day 1) vs Givinostat Co-Administered With Clarithromycin (Day 8); Test type: Superiority; ratio of the Geometric LSmeans = 117.97, 90% CI 2-sided [112.24 to 124.00]

3. Primary Outcome: AUC0-inf of Givinostat, Following Single Doses of the Parent Drug
Description: AUC0-inf=Total AUC extrapolated to infinity, calculated as AUC0-t + Clast/λz, where Clast is the last measurable concentration and λz is the apparent terminal elimination rate constant.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of givinostat.
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 19 | 19
ng.h/mL | 349.25 (20.1) | 411.69 (12.7)
Statistical Analysis 1: Comparison: Givinostat Alone (Day 1) vs Givinostat Co-Administered With Clarithromycin (Day 8); Test type: Superiority; ratio of the Geometric LSmeans = 117.88, 90% CI 2-sided [112.13 to 123.92]

4. Primary Outcome: %AUCextrap of Givinostat, Following Single Doses of the Parent Drug
Description: %AUC0extrap = Percentage of AUC0-∞ due to extrapolation from the time of the last measurable concentration (tlast) to infinity, i.e., residual area, calculated as 100 ·(AUC0-∞ - AUC0-t) / AUC0-∞.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of givinostat
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-∞
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 19 | 19
percentage of AUC0-∞ | 1.28 (23.3) | 1.17 (29.7)

5. Primary Outcome: Tmax of Givinostat, Following Single Doses of the Parent Drug
Description: Tmax =The time of occurrence of maximum observed concentration of Givinostat.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of Givinostat.
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: Pharmacokinetic Analysis Population: subjects enrolled in the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation. Please note that in the combo arm, one of the 20 PK subjects early withdrew from the study before taking the drug combination. This explains why patients analyzed in the combo arm are n=19 and not n=20.
Measure: Median (Full Range); unit: hours
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 20 | 19
hours | 2.00 [1.00 to 4.00] | 1.50 [0.50 to 2.50]

6. Primary Outcome: λz of Givinostat, Following Single Doses of the Parent Drug
Description: λz is the apparent first order elimination rate constant associated with the terminal (log-linear) portion of the concentration versus time curve. The parameter is estimated by linear least square regression analysis using the last three (or more) non- zero concentrations.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of givinostat
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: Pharmacokinetic Analysis Population: subjects enrolled in the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation. Please note that one of the 20 PK subjects early withdrew from the study before taking any study drug. This explains why patients analyzed in each arm are n=19 and not n=20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 19 | 19
1/hour | 0.112 (4.9) | 0.103 (23.2)

7. Primary Outcome: t1/2 of Givinostat, Following Single Doses of the Parent Drug
Description: t1/2 is the apparent terminal elimination half-life, calculated as ln(2)/λz.
  A total of 40 blood samples were collected as follows:
  - Twenty (20) blood samples at pre-dose and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 60 and 72 hours after the administration of givinostat, on Days 1 and 8, for the determination of Givinostat.
Time Frame: In the turn of 72 hours after administration of Givinostat
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Givinostat Alone (Day 1) | Givinostat Co-Administered With Clarithromycin (Day 8)
Number analyzed (Participants) | 19 | 19
hours | 6.18 (4.9) | 6.70 (23.0)

8. Secondary Outcome: Severity of Treatment Emergent Adverse Events (TEAE)
Description: An AE was considered as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily imply a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The period of observation for the collection of medical occurrences extended from the time when the subject gave Informed Consent until the follow-up visit.
Time Frame: Throughout the study and 10-14 days after the EoS (follow-up visit), i.e. up to day 30-34
Population: Pharmacokinetic Analysis Population: subjects enrolled in the study, who provided evaluable pharmacokinetic data for at least one IMP, without deviations affecting pharmacokinetic interpretation. For one of the 20 PK subjects, though, data at day 8 are missing.
Measure: Number; unit: number of events
Groups:
- Givinostat: givinostat 50 mg as oral suspension was administered as a single dose, on Days 1 and 8
- Clarithromycin: Clarithromycin 500 mg immediate-release film-coated tablets (Klacid®) b.i.d. Days 4-7, 9-10
- Total Enrolled: Givinostat 50 mg Day 1 Clarithromycin 500 mg b.i.d. Days 4-7 Clarithromycin 500 mg b.i.d + Givinostat 50 mg Day 8 Clarithromycin 500 mg b.i.d. Days 9-10
Arm/Group | Givinostat | Clarithromycin | Total Enrolled
Number analyzed (Participants) | 20 | 19 | 20
number of events
  mild | 43 | 41 | 43
  moderate | 3 | 0 | 3
  severe | 0 | 0 | 0
  total | 46 | 41 | 46

ADVERSE EVENTS:
Time Frame: Throughout the study and 10-14 days after the End of Study (follow-up visit), i.e. up to day 30-34, all TEAEs, considered related or not related to IMPs, were collected.
Description: End-of-study was defined as the last study procedure on Day 11 or at early discontinuation of subjects administered at least one dose of investigational product.
  Early termination procedures were performed as soon as possible after subject withdrawal, within 10-14 days after last participation of the subject in the study, whenever possible
Arm/Group | Givinostat | Clarithromycin | Total Enrolled
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 16/20 | 16/19 | 16/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Givinostat (N=20) | Clarithromycin (N=19) | Total Enrolled (N=20)
Abdominal pain (Gastrointestinal disorders) | 4 (7) | 4 (7) | 4 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (7) | 4 (5) | 4 (7)
Migraine (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 7 (7) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT05845567/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT05845567/SAP_001.pdf